CLINICAL TRIAL: NCT03915613
Title: Brain Insulin Resistance and Motivation in Mood Disorders
Brief Title: Brain Insulin Resistance in Mood Disorders
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Rodrigo Mansur, Psychiatrist, Assistant Professor of Psychiatry at the University of Toronto, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-5789.0
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Anhedonia; Intranasal Insulin
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Anhedonia | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: Single-dose, randomized, double-blinded, cross-over study (150 participants) wherein study participants will receive a total of two doses (i.e., one insulin, one placebo) with a washout period of 1 week.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin (Experimental): Intranasal insulin will be made prepared from Humulin® R [insulin injection, human biosynthetic (rDNA Origin) REGULAR; 10 mL/vial, manufactured by Eli Lilly]. Each mL contains: 100 units of insulin injection, human biosynthetic (rDNA Origin) REGULAR. Nonmedicinal ingredients contain: glycerol, hydrochloric acid, m-cresol, sodium hydroxide and water for injection.
  Unopened vials should be stored under refrigeration between 2°C and 8°C (36°F to 46°F) until the expiration date; do not freeze; keep away from heat and sunlight. Once punctured (in use), Humulin vials should be stored at room temperature <25°C (<77°F) and discarded after 28 days.
  To obtain a dose Humulin R 160 U / placebo
  * 16 sprays (0.1 mL/spray) are to be given per dose
  * This works out to 16 sprays split between each nostril such that each nostril receives 8 sprays.
  * The sprays will be administered between alternating nostrils
  Interventions: Drug: Humulin R
- Sterile Diluent (Placebo Comparator): Intranasal placebo will be prepared from Eli Lilly's sterile diluent used with Humulin® R (10 mL/vial, manufactured by Eli Lilly). Nonmedicinal ingredients contain: dibasic sodium phosphate, glycerin, liquefied phenol, metacresol, hydrochloric acid, sodium hydroxide and water for injection.
  Unused sterile diluent should be kept at controlled room temperature until the expiration date. The USP defines controlled room temperature as (20° to 25°C [68° to 77°F]), with excursions permitted (15° to 30°C [59° to 86°F]). Once in-use, the sterile diluent vial should be used within 28 days.
  Participants will follow the same dosage, frequency, and administration as Humulin:
  * 16 sprays (0.1 mL/spray) are to be given per dose
  * This works out to 16 sprays split between each nostril such that each nostril receives 8 sprays.
  * The sprays will be administered between alternating nostrils
  Interventions: Drug: Diluent

INTERVENTIONS:
Drug: Humulin R — The investigator and/or designee will instruct the study participant on how the intranasal insulin spray should be administered. Each study participant is to receive a single dose of Humulin R 160 U.
  The nasal spray bottles provide a deliverable volume of 0.1 mL/spray. Humulin R insulin will be sourced as 100 units/mL in a vials of 10 mL from Eli Lilly. 16 sprays in alternating nostrils (8 per nostril) will be administered per dose.
  Arms: Insulin
Drug: Diluent — The investigator and/or designee will instruct the study participant on how the intranasal placebo spray should be administered. Each study participant is to receive a single dose of placebo.
  The nasal spray bottles provide a deliverable volume of 0.1 mL/spray. Diluent will be sourced as 10 mL/vial from Eli Lilly. 16 sprays in alternating nostrils (8 per nostril) will be administered per dose.
  Arms: Sterile Diluent

SUMMARY:
The overarching aim of the study is to determine the role of insulin signaling on the neurobiological substrates subserving anhedonia within individuals with mood disorders (i.e., Bipolar Disorder (BD) and Major Depressive Disorder (MDD)).

Specific aims include:

1. Molecular: Assessment of components of the insulin cascade, as well as of anhedonia and reward-related processes, using a proteomics and gene expression approach;
2. Physiology: Measurement of peripheral sensitivity to insulin and metabolic correlates, including body mass index and dyslipidemia;
3. Neural Circuits: Evaluation of the insulin sensitivity of prefrontal (e.g. prefrontal cortex) and striatal (e.g. nucleus accumbens, ventral tegmental area) networks in the resting-state and during an effort-based decision making test, using acutely administered intranasal insulin and functional magnetic resonance imaging (fMRI);
4. Behavioral: Measurement of willingness to make effort for rewards, as well as of other components of reward response and anhedonia, using validated behavioral tasks and clinical scales (e.g. Snaith-Hamilton Pleasure Scale - SHPS).

This initiative represents a proof-of-concept study that insulin is important to anhedonia, neurocognitive functioning, and behavioural deficits in MDD, representing a novel and safe therapeutic avenue.

DETAILED DESCRIPTION:
Seventy-five adults between the ages of 18 to 50 years with DSM-5 defined MDD or BDI/II, in a depressive episode will be enrolled, in addition to seventy-five age- and sex-matched healthy controls. Enrollment into the study is voluntary. Eligible participants will provide written informed consent. Participants will be enrolled from the outpatient Mood Disorders Psychopharmacology Unit (MDPU), University Health Network (UHN), University of Toronto.

The MDPU case report form will gather information on the participant's course of illness variables. Conventional pharmacological treatments for MDD and BD will be permitted.

Participants will be excluded if they are receiving insulin and/or oral hypoglycemiants; have been diagnosed with possible or probable Alzheimer's Disease, Mild Cognitive Impairment, or any other dementia; have a history of neurological disorder, or evidence of neurologic or other physical illness that could produce cognitive deterioration; have substance use disorder within 3 months before screening or a positive baseline toxicology screen; have a clinically unstable general medical illness; are pregnant or breastfeeding; have MRI contraindications.

The ongoing provision of care is not contingent on enrollment and/or completion of the study protocol. Furthermore, there will be ongoing communication with the participant's primary care provider in regards to their participation in this study.

This is a randomized double-blind, placebo-controlled, cross-over study. The initial visit entails the provision of detailed study information to the patient and obtainment of written informed consent from the participant. The participant will then meet a research team member at a later date for a screening visit. This study requires a total of 3 visits: one screening visit and two fMRI scan visits.

Screening and Baseline Assessment: Subjects will first meet with a staff psychiatrist for a clinical consultation. After obtaining consent and if inclusion criteria are met, a medical comorbidity questionnaire will be administered to screen for concurrent and lifetime medical conditions. Participant's demographic characteristics and current medications, as well as lifetime psychotropic medications received will be recorded. The investigators will also assess dietary intake with the short food frequency questionnaire (SFFQ); smoking, by questioning number of cigarettes smoked per day, age when smoking stated, and quit date, if applicable, to calculate a smoking pack-year history; physical activity using the International Physical Activity Questionnaire (IPAQ); and alcohol and/or substance abuse with the Addiction Severity Index (ASI). In addition, the investigators will assess demographics, socioeconomic status, medical history, and family psychiatric history; childhood trauma history with the Childhood Trauma Questionnaire (CTQ) will also be assessed. Participants will also be asked to complete an MRI screening questionnaire to ensure that they have no contraindications. The following self-reported measures will be carried out: Perceived Deficits Questionnaire-Depression (PDQ-D), Sheehan Disability Scale (SDS), UCLA life Stress (Episodic), DeJong Gierveld Loneliness Scale, Pittsburg Sleep Quality Index (PSQI), Social and Occupational Functioning Assessment Scale (SOFAS). Participants will be required to complete a urine drug screen. Female participants will be asked to do blood work to confirm they are not pregnant.

Physiological Assessment: Anthropometric (i.e. BMI, waist-hip ratio) and metabolic measurements (i.e. fasting glucose, fasting insulin, glycated hemoglobin, lipids and HOMA-IR) will be completed at each study visit.

Behavioral assessment: These tasks are simple, user-friendly tools that provide an opportunity, when used in conjunction with the most widely used questionnaires, to gain novel insights on reward behaviors in mood disorders.

1. The primary behavioral measurement will be effort-based decision-making, assessed using the Effort-Expenditure for Rewards Task (EEfRT), which will be done in a fMRI paradigm.
2. Assessments will include the validated anhedonia scale Snaith-Hamilton Pleasure Scale (SHPS), and the mood questionnaires Montgomery-Åsberg Depression Rating Scale (MADRS), and Young Mania Rating Scale (YMRS) during each study visit.

Neural Circuits Assessment: A promising tool to study the effect of insulin on CNS is intranasal insulin, which is delivered directly into the brain, without relevant effects on peripheral glucose. A single dose of intranasal insulin has been shown to influence brain activation, increasing regional perfusion and functional connectivity between the hippocampus and the PFC. Acute administration of intranasal in randomized, placebo-controlled, cross-over designs has been previously used to determine regional responses to insulin in the resting-state or during tasks.

After screening and baseline assessment, participants will receive a crossover treatment assignment of either insulin or diluent followed by an MRI scan, with a washout period of 1 week. Therefore, participants will receive a total of 2 MRI scans throughout the course of the study- one following the first treatment, and one following the second treatment. The subsample will be enriched for the presence of self-reported anhedonia, using a score of greater than 2 on the SHPS as a cut-off, which provides the best discrimination between "normal" and "abnormal" level of hedonic tone. This subsample will also have equal representation of normal weight and obese participants. Imaging procedures will be done in collaboration with the Centre for Addiction and Mental Health (CAMH). CAMH is Canada's largest mental health teaching hospital and one of the world's leading research centres in its field. CAMH is fully affiliated with the University of Toronto and is a Pan American Health Organization/World Health Organization Collaborating Centre.

To proxy insulin activity within pre-selected brain regions, the investigators will use a provocation paradigm, involving the administration of exogenous intranasal insulin, based on the published work of other research groups. Activation of brain regions will be assessed during the resting state and task-based reward paradigm (i.e. EEfRT), following an intranasal administration of either 160 units of intranasal insulin or diluent (insulin and placebo will be prepared as nasal sprays), in a randomized, double-blinded, cross-over design. A hypothesis-driven region of interest approach will be used to investigate initially the striatum and the medial PFC (mPFC). Willingness to make effort for rewards will be measured with the EEfRT.

Imaging procedures will be started with a safety monitoring for glucose and cardiovascular vital signs. An insulin/placebo spray will be administered intranasally and, within 30 min, fMRI measurement will be performed. Venous blood samples, for determination of plasma glucose and insulin concentrations, will be obtained at the time of the insulin/placebo spray administration and immediately after the scan. The 2 scans for each individuals will be acquired on the same scanner. Subjects will be scanned using a 3.0-Tesla Signa HDx scanner with an 8-channel phased-array receiver coil (GE Healthcare, Milwaukee, Wisconsin) consisting of a structural and functional neuroimaging, comprising:

1. Whole-brain 3-D T1-weighted Inversion-Recovery prepared Fast Spoiled Gradient-Echo (IR-FSPGR) anatomical scan with the following parameters: (TI/TR/TE = 450/8/3 ms, matrix size 256 × 256, field of view 22 × 22 cm, slice thickness = 1 mm, and flip angle = 15°)
2. Whole-brain, T2*-weighted BOLD echo planar imaging (EPI) during awake resting state with the following parameters: (TR/TE = 2000/30 ms, 3.5 x 3.5 x 3.5 mm voxel size, field of view 24x24 cm, 39 slices, slice thickness 3.5 mm, matrix size 64x64, number of frames = 405, flip angle = 70°)),
3. Three runs of whole-brain, T2*-weighted BOLD EPI series during task-based reward paradigm with the same parameters as in ii.

ELIGIBILITY:
Inclusion criteria (patients):

1. Age 18-60
2. DSM-5 defined MDD/BD and a total score ≥20 on the Montgomery-Åsberg Depression Rating Scale (MADRS) and no history of dementia or intellectual disability
3. A written, voluntary informed consent prior to study enrollment

Exclusion criteria (patients):

1. Use of insulin and/or oral hypoglycemiants, due to its confounding effects
2. Diagnosis of possible or probable AD, MCI, or any other dementia
3. History of neurological disorder, or evidence of neurologic or other physical illness that could produce cognitive deterioration
4. Substance use disorder within 3 months before screening or a positive baseline toxicology screen
5. Presence of clinically unstable general medical illness
6. Pregnancy or breastfeeding
7. MRI contraindications

Inclusion criteria (healthy controls):

1. Age 18-60
2. A written, voluntary informed consent prior to study enrollment

Exclusion criteria (healthy controls):

1. Use of insulin and/or oral hypoglycemiants, due to its confounding effects
2. Presence of any current or lifetime psychiatric or neurological conditions
3. Substance use disorder within 3 months before screening or a positive baseline toxicology screen
4. Presence of clinically unstable general medical illness
5. Pregnancy or breastfeeding
6. MRI contraindications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-10-05 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Effort-Expenditure for Rewards Task (EEfRT) | 2 weeks
  Score from the end of each treatment phase.

SECONDARY OUTCOMES:
Young Mania Rating Scale (YMRS) | 2 weeks
  Scale that assesses manic symptoms. The scale has 11 items and is based on the patient's subjective report of his/her clinical condition over the previous 48 hours. Additional information is based upon clinical observations made during the course of the clinical interview. Each item assesses a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Typical YMRS baseline scores can vary a lot and they depend on the patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2). A higher total score is indicative of worse outcome.
Montgomery-Asberg Depression Scale (MADRS) | 2 weeks
  Scale that assesses depressive symptoms. The scale has 10 items and is based on the patient's subjective report of his/her clinical condition over the previous 7 days. Additional information is based upon clinical observations made during the course of the clinical interview. Each item assesses a severity rating. All items that are graded on a 0 to 6 scale. The overall MADRS score ranges from 0-60. Higher scores are indicative of more severe depression.Usual cutoff points are: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; >34 - severe depression.
Snaith-Hamilton Pleasure Scale (SHAPS) | 2 weeks
  The SHAPS is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Thus, the final score ranges from 0 to 14 and higher scores are indicative of greater anhedonia.
Perceived Deficits Questionnaire-Depression (PDQ-D) | 2 weeks
  The PDQ-D is a 20-item, patient-reported questionnaire with a 7-day recall period. Scores for four subscales of the PDQ-D (attention/concentration, retrospective memory, prospective memory, and planning/organization) are computed based on responses to five items in each subscale. All 20 items use the same 5-point ordinal categorical response scale to reflect the frequency of experiencing a specific cognitive problem. Scores for each of the four measured subscales are calculated by assigning a value of 0 ("never in the past 7 days"), 1 ("rarely - once or twice"), 2 ("sometimes - 3-5 times"), 3 ("often - about once a day"), or 4 ("very often - more than once a day") to each item, then summing the five items of that subscale, to produce a score ranging from 0 to 20. A total global score for overall cognitive dysfunction (range 0-80) is calculated by summing the four subscale scores. Higher scores for each subscale and for the total score indicate greater perceived cognitive dysfunction.
Sheehan Disability Scale (SDS) | 2 weeks
  The SDS is a brief 3-item self-report tool that assesses functional impairment in work/school, social life, and family life on a 10-point visual analog scale. Each subdomain has a rating from 0-10 and can be added up to determine the total score. Scores equal to or greater than 5 on each subdomain indicate significant functional impairment and as such, higher total scores are indicative of this as well (Total score 0-30; 0=unimpaired, 30= highly impaired).
The DeJong Gierveld Loneliness Scale | 2 weeks
  The DeJong Gierveld Loneliness Scale is a 6-item scale, wherein three statements are made about 'emotional loneliness' and three about 'social loneliness'. There are negatively (items 1-3) and positively (items 4-6) worded items. On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Therefore, on questions 4-6, score Yes=0, More or less=1, and No=1. This gives a possible range of scores from 0 to 6, which can be read as follows: 0= least lonely; 6= most lonely.
International Physical Activity Questionnaire (IPAQ) | 2 weeks
  The IPAQ comprises a set of 4 questionnaires. Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks
  The PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by summing the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Social and Occupational Functioning Assessment Scale (SOFAS) | 2 weeks
  The SOFAS is a scale that focuses exclusively on the individual's level of social and occupational functioning and is not directly influenced by the overall severity of the individual's psychological symptoms. The SOFAS is used to rate functioning for the current period (i.e., the level of functioning at the time of the evaluation) on a scale from 1-100. A higher score is indicative of greater social and occupational functioning.
  The interviewer must consider social and occupational functioning on a continuum from excellent functioning to grossly impaired functioning, including impairments in functioning due to physical limitations, as well as those due to mental impairments. To be counted, impairment must be a direct consequence of mental and physical health problems; the effects of lack of opportunity and other environmental limitations are not to be considered.
Digit Symbol Substitution Test (DSST) | 2 weeks
  Neurocognitive task. Score from the end of each treatment phase.
Rey Auditory Verbal Learning Test (RAVLT) | 2 weeks
  Neurocognitive task. Score from the end of each treatment phase.
Trail Making Test A/B (TMT A/B) | 2 weeks
  Neurocognitive task. Score from the end of each treatment phase.

OTHER OUTCOMES:
Height (ft) | 2 weeks
  Height measured at first visit only.
Weight (kg) | 2 weeks
  Weight measured at each visit.
Blood Pressure (mmHG) | 2 weeks
  Blood pressure measured at each visit.
Heart Rate (Bpm) | 2 weeks
  Heart rate measured at each visit.
Waist/hip circumference (cm) | 2 weeks
  Waist/hip circumference measured at each visit.
Childhood Trauma Questionnaire- CTQ | 2 weeks
  The CTQ is a brief survey of six early traumatic experiences (death, divorce, violence, sexual abuse, illness or other), and assesses individual's understanding of their childhood trauma. The scores for each subdomain are as follows:
  Emotional Abuse: None=5-8; Low=9-12; Moderate=13-15; Severe=16+ Physical Abuse: None=5-7; Low=8-9; Moderate=10-12; Severe=13+ Sexual Abuse: None=5; Low=6-7; Moderate=8-12; Severe=13+ Emotional Neglect: None=5-9; Low=10-14; Moderate=15-17; Severe=18+ Physical Neglect: None=5-7; Low=8-9; Moderate=10-12; Severe=13+ Higher scores in each of the subdomains indicate greater (i.e., more severe) trauma.
UCLA Episodic Life Stress Interview | 2 weeks
  The UCLA Episodic Life Stress Interview is the assessment of episodic stressors over the past 6 months. Interviewers obtain detailed information regarding the nature and date of each event, and the circumstances in which each event occurred (e.g., whether the event was expected or unexpected, how long it continued, whether the person had previous experience with the event, and consequences of the event). Based on this information, the interviewer makes am objective rating of how much impact the event would have on a typical person under similar circumstances. Objective ratings of event severity range from 1 (no impact) to 5 (extremely severe impact). The interviewer also rates the extent to which each event was dependent on the participant's behavior, using a 1 (entirely independent) to 5 (entirely dependent) scale. In both ratings, higher scores are indicative of greater stress.
Short Food Frequency Questionnaire (SFFQ) | weeks
  The SFFQ is a method of collecting the participant's dietary intake on a weekly basis.
Addiction Severity Index (ASI) | 2 weeks
  The ASI is a semi-structured interview designed to address seven potential problem areas in substance-abusing patients: medical status, employment and support, drug use, alcohol use, legal status, family/social status, and psychiatric status. A skilled interviewer will gather information on recent (past 30 days) and lifetime problems in all of the problem areas. The ASI provides an overview of problems related to substance, rather than focusing on any single area.
  The severity ratings are interviewer estimates of the patient's need for additional treatment in each area. The scales range from 0 (no treatment necessary) to 9 (treatment needed to intervene in life-threatening situation). Each rating is based upon the patient's history of problem symptoms, present condition and subjective assessment of his/her treatment needs in a given area.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT03915613/Prot_SAP_002.pdf
  • Informed Consent Form: Patient Participants (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03915613/ICF_003.pdf
  • Informed Consent Form: Healthy Participants (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03915613/ICF_004.pdf